CLINICAL TRIAL: NCT02197533
Title: Educating Patients on Management of Overactive Bladder: Written Versus Verbal Instructions
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Unity Health Toronto (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 14-213
Record Dates: First submitted 2014-07-21; First posted 2014-07-22 (Estimated); Last update posted 2019-12-04 (Actual); Status verified 2019-12

CONDITIONS: Overactive Bladder
MeSH Terms: conditions — Urinary Bladder, Overactive

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Written list (Experimental): Patients in the intervention group will receive both verbal information and a written supplement (Appendix 1), produced during the discussion by CM or a fellow (not the individual who obtained consent), on treatment recommendations for OAB. They will leave clinic with this written list of recommendations and will be able to take it home with them.
  Interventions: Other: Written List
- Control (No Intervention): Patients in the control group will receive the same verbal information on the treatment recommendations for OAB, however, these patients will not receive the written list of management strategies for their condition.

INTERVENTIONS:
Other: Written List — Written list of seven management strategies for OAB to be produced during verbal discussion about management.
  Arms: Written list

SUMMARY:
Background: Overactive bladder (OAB) is a common condition among postmenopausal women, requiring a multifaceted treatment approach that requires patient retention of information given to them in clinic. Recall of recommendations is a key component of compliance. Supplemental educational tools such as handouts and audiovisual information have been investigated for their ability to improve patients' recall of information and increase satisfaction with the clinical encounter.

Objective: To determine if a written list of seven management strategies for overactive bladder leads to improved immediate and delayed recall of these recommendations in postmenopausal women presenting with OAB compared to a traditional verbal discussion.

Methods: In this single-blind, randomized controlled trial, patients' immediate and delayed (2-week) recall of seven OAB management strategies will be compared between two groups. The intervention group will receive a handwritten list during their verbal discussion of OAB treatment while the control group will receive standard care (verbal discussion only). Immediate and delayed recall will be assessed by a member of the study team who has been blinded to participants' group assignments.

Results: The results of this study may guide clinicians in the most effective mode of providing treatment recommendations to post-menopausal patients with OAB.

ELIGIBILITY:
Inclusion Criteria:

* New diagnosis of overactive bladder
* post-menopausal

Exclusion Criteria:

* Pre-existing diagnosis of dementia or other cognitive disorders
* Patients with mixed incontinence
* Non-English speaking
* Patients with contraindications to taking vaginal estrogen or anticholinergic medications

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2014-07; Primary Completion 2018-01-31 (Actual); Study Completion 2019-09-01 (Actual)

PRIMARY OUTCOMES:
Recall | 0 and 2 weeks
  Mean number of treatment strategies recalled (scored out of seven) immediately and two weeks after the clinic appointment.

CONTACTS AND LOCATIONS:
Overall Officials: Colleen McDermott, MD, MSc, FRSCS, Principal Investigator — Unity Health Toronto
Locations (1):
- St. Michael's Hospital, Toronto, Ontario, Canada